CLINICAL TRIAL: NCT04328155
Title: The Effectiveness of Different Electrophysical Agents on Hamstring Muscles Flexibility in Healthy Individuals
Brief Title: Effects of Different Electrophysical Agents in Hamstring Muscles Flexibility of Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Nur OYMAK SOYSAL, Lecturar, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26.06.2018/13
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-03

CONDITIONS: Flexibility; Hamstring Muscles
Keywords: electrophysical agents; stretching exercises; hamstring muscles

STUDY DESIGN:
Intervention Model Description: parallel assingment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hotpack Group (Experimental): Group I (15 subjects) received 18 sessions hotpack to hamstring muscles and self stretching exercise3 times per week.
  Interventions: Procedure: Hotpack Group
- Infrared Group (Experimental): Group II (15 subjects) received 18 sessions infrared to hamstring muscles and self stretching exercise3 times per week.
  Interventions: Procedure: Infrared Group
- Ultrasound Group (Experimental): Group III (15 subjects) received 18 sessions ultrasound to hamstring muscles and self stretching exercise 3 times per week.
  Interventions: Procedure: Ultrasound Group
- Control (Active Comparator): Group IV (15 subjects) received 18 sessions self stretching exercise 3 times per week.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Hotpack Group — Hotpack Group received 20 minutes hotpack to hamstring muscles region at prone position and participants stretched the hamstring muscles at supine position.Self stretching hamstring exercise was done by straight leg lifting using a band three times for 15 seconds .
  Arms: Hotpack Group
Procedure: Infrared Group — Infrared Group received 20 minutes infrared to hamstring muscles region at prone position and participants stretchted the hamstring muscles at supine position.Self stretching hamstring exercise was done by straight leg lifting using a band three times for 15. seconds .
  Arms: Infrared Group
Procedure: Ultrasound Group — Ultrasound Group received 5 minutes 1 M-Hz, 1,5 watt/cm2 ultrasound therapy to hamstring muscles region at prone position and participants stretched the hamstring muscles at supine position.Self stretching hamstring exercise was done by straight leg lifting using a band three times for 15 seconds .
  Arms: Ultrasound Group
Procedure: Control — Control Group participants stretched the hamstring muscles at supine position.Self stretching hamstring exercise was done by straight leg lifting using a band three times for 15 seconds .
  Arms: Control

SUMMARY:
Sixty healthy individuals will be randomised into four groups. Group I (15 subjects) will be applied hotpacks, Group II (15 subjects) will be applied infrared, Group III will be applied ultrasound to hamstring muscles for 18 sessions 3 times per week and the subjects will do hamstring self stretching exercise 3 times for 15 seconds. Group IV will only do self stretching exercises.

Outcome measures are Range of Motion and hamstring flexibility. Measurements will record before and after the end of the treatment.

DETAILED DESCRIPTION:
Inclusion criteria for the study are; being student of Saraykoy Vocational School, Active knee extension degree must be lower than 60 when the hip flexed to 90 degree. Exclusion criteria are; undergoingsurgery for knee pathologies, having a systemic and inflammatory disease targeting this region, having a knee disorder, pregnancy, malignancy, doing regularly another exercise programme. According to our criteria 60 participants will be randomised into four groups. Group 1 will receive 20 minutes hotpacks and will do hamstring self stretching exercise 3 times for 15 seconds. Participants will do self stretching hamstring exercise at supine position lying and they will use a band for stretching. Group II will receive 20 minutes infrared at prone position and will do self stretching exercise 3 times for 15 seconds. Participants will do self stretching hamstring exercise at supine position lying and they will use a band for stretching.

Group III will receive 5 minutes 1MHz ultrasound therapy and will do self stretching exercise for 18 sessions 3 times per week. Participants will do self stretching hamstring exercise at supine position lying and they will use a band for stretching 3 times for 15 seconds. Group IV will do only hamstring self stretching exercise therapy for 18 sessions 3 times per week. Participants will do self stretching hamstring exercise at supine position lying and they will use a band for stretching 3 times for 15 seconds. Outcome measures are Range of Motion and hamstring flexibility. Range of Motion will be assed by using universal goniometer for knee and hip joints. Hamstring flexibility will be assed with active knee extension test by using universal goniometer. All measurements will done 3 times and average of scores will be taken. Outcomes will be recorded before and after the end of the treatment. All assessments were made by the same researcher before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being Student in Saraykoy Vocational School
* Having Active Knee Extension degree lower than 60

Exclusion Criteria:

* undergoing surgical operation for knee pathologies
* history of trauma involving knee joint region
* having a systemic and inflammatory disease targeting this region
* pregnancy
* malignancy
* doing another exercise programme

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2021-08-28 (Estimated)

PRIMARY OUTCOMES:
Changes of ROM | baseline, after 6 weeks
  Range of motion was measured by universal goniometer. Knee flexion and extension, Hip flexion, extension, external and internal rotation was measured
Hamstring Flexibility | baseline, after 6 weeks
  Hamstring Flexibility was measured by universal goniometer by using active knee extension test.

CONTACTS AND LOCATIONS:
Overall Officials: Atiye KAŞ ÖZDEMİR, Msc, Study Chair — Sarayköy Vocational School Turan Mah. Jeotermal Sok. No:1 Sarayköy, Denizli; Ummuhan BAŞ ASLAN, Prof .Dr., Study Chair — Pamukkale Univercity 20070 Kınıklı Denizli, Turkey; Merve Bergin KORKMAZ, DR., Study Chair — Denizli State Hospital 20040 Denizli, Turkey
Locations (1):
- Sarayköy Vocational School, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because there is no web site to share my data

REFERENCES:
- [Result] Sadler SG, Spink MJ, Ho A, De Jonge XJ, Chuter VH. Restriction in lateral bending range of motion, lumbar lordosis, and hamstring flexibility predicts the development of low back pain: a systematic review of prospective cohort studies. BMC Musculoskelet Disord. 2017 May 5;18(1):179. doi: 10.1186/s12891-017-1534-0. PMID 28476110
- [Result] Burke DG, Holt LE, Rasmussen R, MacKinnon NC, Vossen JF, Pelham TW. Effects of Hot or Cold Water Immersion and Modified Proprioceptive Neuromuscular Facilitation Flexibility Exercise on Hamstring Length. J Athl Train. 2001 Mar;36(1):16-19. PMID 12937509
- [Result] Brodowicz GR, Welsh R, Wallis J. Comparison of stretching with ice, stretching with heat, or stretching alone on hamstring flexibility. J Athl Train. 1996 Oct;31(4):324-7. PMID 16558418